CLINICAL TRIAL: NCT06154668
Title: Phenotypic, Functional, Metabolic and Transcriptomic Profiling of Circulating Immune Cells to Uncover Response Signatures to Anti-PD1 Immunotherapy in Melanoma Patients
Brief Title: Profiling of Circulating Immune Cells to Uncover Response Signatures to Anti-PD1 Immunotherapy in Melanoma Patients
Acronym: PHENOMENAL
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Etablissement Français du Sang (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC23.0280; 2023-A01722-43 (Other: ID RCB)
Record Dates: First submitted 2023-11-23; First posted 2023-12-04 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Cohort #A: monotherapy anti-PD1 first line
- Cohort #B: monotherapy anti-PD1 second line
- Cohort #C: monotherapy anti-PD1 adjuvant
- Cohort #D: combotherapy anti-PD1/CTLA-4 first line
- Cohort #E: untreated stage I and II melanoma patient

SUMMARY:
Despite being standard of care, there are still many medical requirements related to immune checkpoint blocker based therapies such as identify patients susceptible to respond with the less adverse events, evaluate the clinical benefit of adjuvant treatment /risk of relapse and design new strategies for non-responder patients.

Thus, this project aims at understanding the impact of anti-PD1 on the immune system through investigation of the phenotypic, functional, metabolic and transcriptomic profiles of circulating DC subsets and effectors in response to anti-PD1 therapy in melanoma patients.

The primary objective of the study is to identify the biomarkers of response to anti-PD1 according to the type of patient before the start of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patient with histologically confirmed melanoma (stage I, II, III or IV based on AJCC classification)
* Able to sign the informed collection consent for the retrospective part or to express their non-opposition to the research for the prospective part of the study

Exclusion Criteria:

* Subject under guardianship or subject deprived of freedom
* Persons benefiting from special protection (as defined in Articles L1121-5 and L1121-8 of the Public Health Code): minors, pregnant or breastfeeding women, adults protected by law (under guardianship, curatorship or deprived of liberty) and persons hospitalized without their consent (as defined in Articles L3212-1 and L3212-3 of the Public Health Code).
* ocular melanoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with unresectable (stage III) or metastatic (stage IV) melanoma, followed at CHU Grenoble - Alpes in Dermatology deparment for diagnosis, follow-up or recurrence of melanoma, and treated with immune checkpoint blocker in curative or adjuvant setting.
Sampling Method: Probability Sample
Enrollment: 707 (Estimated)
Dates: Start 2024-01-17 (Actual); Primary Completion 2030-01 (Estimated); Study Completion 2031-01 (Estimated)

PRIMARY OUTCOMES:
Identification of biomarkers of response to anti6PD1 according to the type of patient before the start of treatment | 6 months
  response to treatment according to immunological parameters at T0 between patients responding (R), stable (SD) and non-responding (NR) to treatment

SECONDARY OUTCOMES:
identification of early biomarkers predictive of the response to anti-PD1 | at each time point (3, 4 or 6 weeks)
  comparison of immunological parameters according to the type of patients (R, SD and NR) for each time point

CONTACTS AND LOCATIONS:
Overall Officials: Julie Charles, MD, PhD, Principal Investigator — CHU Grenoble Alpes
Locations (1):
- CHU Grenoble Alpes, Grenoble, France